CLINICAL TRIAL: NCT03446755
Title: The Use of an Intrauterine Balloon in Preventing Adhesion Recurrence After Hysteroscopic Adhesiolysis: a Feasibility Study.
Brief Title: Use of an Intra Uterine Balloon to Prevent Recurrent Adhesions (REpAIR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: B670201733915
Record Dates: First submitted 2018-01-24; First posted 2018-02-27 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Adhesion; Uterus, Internal
Keywords: antiadhesion treatment; Asherman's syndrome; hysteroscopic adhesiolysis; intrauterine adhesions; intrauterine balloon
MeSH Terms: conditions — Tissue Adhesions; Gynatresia

STUDY DESIGN:
Intervention Model Description: To evaluate the feasibility of a hearth shaped intrauterine balloon as antiadhesion method subsequent to a hysteroscopic adhesiolysis in terms of surgeon's and patient's experience.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intrauterine balloon (Cook medical) (Experimental): Insertion of a hearth shaped intrauterine balloon immediately after hysteroscopic adhesiolysis and left in place for 7 days under antibiotic prophylaxis.
  Interventions: Device: intra uterine Cook balloon

INTERVENTIONS:
Device: intra uterine Cook balloon — Insertion of a hearth shaped intrauterine balloon immediately after hysteroscopic adhesiolysis and left in place for 7 days under antibiotic prophylaxis.

SUMMARY:
Patients suffering of subfertility as a consequence of intrauterine adhesions could be treated with hysteroscopic adhesiolysis. Adhesion recurrence may occur postoperative. An intrauterine balloon, inserted after hysteroscopic adhesiolysis, may prevent adhesion reformation.

A Foley catheter can serve for this purpose, but its not ideal. COOK medical® developed a hearth shaped intrauterine balloon to reduce bleeding after intrauterine surgery.

We aimed to perform a pilot study of 10 procedures with insertion of a hearth shaped intrauterine balloon as antiadhesion method subsequent to a hysteroscopic adhesiolysis, to study its feasibility in terms of surgeon's and patient's experience.

ELIGIBILITY:
Inclusion Criteria:

* patients with intra uterine adhesions scheduled for hysteroscopic adhesiolysis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female patients will be included
Enrollment: 10 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
The number of recurrent adhesions after adhesiolysis | 5-10 weeks after adhesiolysis
The number of complications after adhesiolysis | 5-10 weeks after adhesiolysis

SECONDARY OUTCOMES:
Pain after placement of the intra uterine balloon | 1 to 6 days after adhesiolysis
  via Visual Analogue Scale (VAS scale). The patient has to indicate her pain score from 0 (no pain) to 10 (worst pain ever).
Complications after placement of the intra uterine balloon | 1 to 6 days after adhesiolysis
Pain at the time of the removal of the intra uterine balloon | 6 days after adhesiolysis
  via Visual Analogue Scale (VAS scale). The patient has to indicate her pain score from 0 (no pain) to 10 (worst pain ever).
Patient Satisfaction after removal of the intra uterine balloon | 6 days after adhesiolysis
  Via questionnaire
Malaise after placement of the intra uterine balloon | 6 days after adhesiolysis
  Via questionnaire
Daily functioning after placement of the intra uterine balloon (absence from work, impact on work productivity, impact on household, physical activity, daily life) | 6 days after adhesiolysis
  Via questionnaire and via via Visual Analogue Scale (VAS scale). The patient has to indicate her daily functioning from 0 (the balloon had no influence on my daily function) to 10 (because of the balloon I couldn't do anything of my daily work).
The ease of inserting the intra uterine balloon | once at the time of the surgical procedure (adhesiolysis). This is day 0 of the study
  Via questionnaire
The ease of removing the intra uterine balloon | 6 days after adhesiolysis
  Via questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Wessel S, Wauters L, Weyers S, Hamerlynck T. The use of an intrauterine balloon in preventing adhesion recurrence after hysteroscopic adhesiolysis: a feasibility study. J Obstet Gynaecol. 2022 Nov;42(8):3720-3724. doi: 10.1080/01443615.2022.2158320. Epub 2022 Dec 21. PMID 36541390